CLINICAL TRIAL: NCT06256627
Title: A Multicenter, Single Arm Clinical Study on the Efficacy and Safety of the "ITIVA" Protocol in Patients With Complete Remission of AML at Initial Diagnosis
Brief Title: The Maintenance Treatment of "ITIVA" in AML Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022-548-002
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2023-08

CONDITIONS: Acute Myeloid Leukemia; Maintenance Treatment; Minor Residue Disease; Interferon-α-1b; Interleukin-2; Thalidomide; Venentoclax; Azacitidine
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Interleukin-2; Thalidomide; Azacitidine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Analyzing the effect of "IFN-α- 1b, il-2, and thalidomide" on negative conversion rate of MRD . (Active Comparator): Analyzing the effect of "interference'- α- 1b, interleukin-2, and thalidomide" on negative conversion rate of MRD in AML patients who have obtained CR or CRi but are MRD positive after routine induction and consolidation chemotherapy
  Interventions: Drug: recombinant human interference'- α- 1b, interleukin-2, thalidomide, Venentoclax and Azacitidine
- To evaluate whether the "ITIVA" regimen as maintenance treatment can improveRFS in AML patients (Active Comparator): To evaluate whether the combination of "recombinant human interference'- α- 1b, interleukin-2, and thalidomide", Venentoclax and Azacitidine triple alternative maintenance treatment can improve relapse free survival (RFS) in AML patients who have achieved CR or CRi through conventional induction and consolidation chemotherapy
  Interventions: Drug: recombinant human interference'- α- 1b, interleukin-2, thalidomide, Venentoclax and Azacitidine

INTERVENTIONS:
Drug: recombinant human interference'- α- 1b, interleukin-2, thalidomide, Venentoclax and Azacitidine — Patients in arm1 were randomly divided into two groups, namely the " interference'- α- 1b, interleukin-2, thalidomide" treatment group and the "VA" treatment group. After receiving a two cycle protocol, patients were evaluated for the endpoint of the trial and their MRD conversion rate was calculated.
  Patients in arm2 will receive triple maintenance treatment, completing three alternative regimens into one cycle. The regimen maintenance treatment will be maintained for a total of 8 cycles. Each medication regimen takes 28 days as a cycle. The number of days administered per cycle can be adjusted based on the patient's blood count.

SUMMARY:
We apply for this clinical study to evaluate the efficacy of "combined recombinant human interference'- α- 1b, interleukin-2, and thalidomide" regimen in obtaining MRD positive AML patients in CR,as well as the efficacy of the "Venentoclax and azacitidine" regimen and the "combined recombinant human interference'- α- 1b, interleukin-2, and thalidomide" regimen in alternately maintaining the treatment of MRD negative AML patients. The study included two cohorts. The first cohort consisted of AML patients who obtained CR or CRi but MRD positive after induction chemotherapy and consolidation chemotherapy. They were randomly given two cycles of "recombinant human interference'- α- 1b, interleukin-2, and thalidomide" or "VA" regimen treatment, and the MRD conversion rates of the two groups were analyzed. In the second cohort , after induction chemotherapy and consolidation chemotherapy, AML patients with CR or CRi and negative MRD were obtained, and were given "recombinant human interference'- α- 1b, interleukin-2, and thalidomide", Venentoclax and Azacitidine triple alternative maintenance treatment, to analyze the impact of maintenance treatment scheme on long-term survival of aml patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, ≥ 14 years old.
2. According to the WHO (2016) diagnostic criteria, the diagnosis of newly diagnosed AML is met (excluding APL).
3. After conventional induction and chemotherapy with at least two consolidation schemes (at least one cycle of the scheme containing medium dose or above of Cytarabine, or the scheme of "vinecla combined with Azacitidine" gets remission, and continues to use the scheme to consolidate at least 6-8 cycles), CR or CRI can be achieved.
4. <6 months from the last chemotherapy.
5. Having sufficient organ functions: creatinine clearance rate ≥ 30 mL/min; Bilirubin<3.0 × Upper limit of normal value (ULN) (sufficient liver function level); Platelets ≥ 50 × 10^9/L; Neutrophil count ≥ 1 × 10^9/L in granulocyte stimulated hematopoietic therapy
6. Whole body functional state score (ECOG) 0-2 points
7. The subjects are willing and able to follow the process required by this protocol.

Exclusion Criteria:

1. Have a history of APL.
2. Morphologically recurrent or refractory AML patients.
3. Previous history of prodromal hematological diseases or treatment-related AML.
4. MRD positive patients are scheduled to undergo allogeneic hematopoietic stem cell transplantation within one month. Patients with negative MRD are scheduled to undergo allogeneic hematopoietic stem cell transplantation within 6 months. Patients who have previously received allogeneic hematopoietic stem cell transplantation.
5. There is a history of AML active central nervous system involvement.
6. HIV infected patients.
7. Uncontrolled infection.
8. Merge New York Heart Association>Level 2 Cardiovascular Dysfunction Status. Level 2 is defined as heart disease where the subject feels comfortable during rest, but regular physical activity can lead to fatigue, palpitations, breathing difficulties, or angina.
9. With chronic Respiratory disease, continuous oxygen inhalation is required, with major medical history of kidney, nerve, spirit, endocrine, metabolism, immunity, liver, cardiovascular disease, or with any other medical condition that the investigator believes will adversely affect his/her participation in this study.
10. Complicated with Malabsorption syndrome or other diseases that hinder the administration of drugs through the intestinal route.
11. Evidence of other clinically significant uncontrollable systemic infections (viruses, bacteria, or fungi) that require treatment.
12. There are mental illnesses/social situations that may affect research compliance.
13. History of merging other malignant tumors under treatment
14. There is a clinically significant medical history or any other reason that the researcher believes will hinder the subject's participation in this study, or make the subject unsuitable for receiving the study drug.
15. There is a history of allergic reactions or significant sensitivity to the ingredients of the investigational drug (and its excipients) and/or other similar products.
16. The subjects are not allowed to receive other anti AML treatments. Non tumor disease treatment drugs can continue to be used.
17. Female subjects with Fertility need to take contraceptive measures.
18. There have been venous or arterial thromboembolic events within the past 6 months.
19. Other researchers believe that it is not suitable for enrollment.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2023-07-11 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
the negative MRD conversion rate of AML patients and whether the combination of triple maintenance treatment can improve relapse free survival (RFS) in AML patients | 2 years
  To evaluate the negative MRD conversion rate of AML patients after "interference'- α- 1b, interleukin-2, and thalidomide" treatment and whether triple maintenance treatment can improve relapse free survival (RFS) in AML patients who have achieved CR or CRi through conventional induction and consolidation chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Xudong None Wei, Doctor/Professor, Principal Investigator — Cancer Hospital of Henan Province
Locations (1):
- The Affiliated Cancer Hospital of Zhengzhou University and Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided